CLINICAL TRIAL: NCT00491647
Title: Time Perception Deficits and Behaviors of Children and Adolescents With Attention-Deficit/Hyperactivity Disorder
Brief Title: Time Perception Deficits and Attention-Deficit/Hyperactivity Disorder
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 9561703011
Record Dates: First submitted 2007-06-23; First posted 2007-06-26 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2008-09

CONDITIONS: Attention-deficit/Hyperactivity Disorder
Keywords: ADHD, time perception, treatments
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background: Literature has documented that children with attention-deficit/ hyperactivity disorder (ADHD) have difficulties in time management by manifesting with difficulties making plans, organizing tasks and activities, and awaiting their turns. However, the studies regarding time perception have been few as compared to those of neuropsychological measures and there is no information about this topic in Chinese population. In view of this, we will conduct a study to investigate the clinical and treatment aspects of time perception among children and adolescent with ADHD.

Specific Aims:

1. to examine the developmental and gender effect on the performance in time perception;
2. to explore the deficit in time estimation, time discrimination, and time reproduction in children and adolescents with ADHD as compared to normal controls;
3. to identify the association between ADHD symptoms and performance in time perception tasks; and
4. to investigate the efficacy of MPH on the time perception measures among children and adolescents with ADHD; Subjects and Methods: This protocol consists of two studies. First, we will recruit 100 patients with DSM-IV ADHD, aged 9 to 16 years, and 100 school controls. They and their parents will receive K-SADS-E interviews. All of them will have complete assessments of time estimation, time discrimination, and time reproduction. Their parents also report on SNAP-IV and CPRS-R:S. The 2nd assessments will be performed 3 months later after the subjects received treatment at outpatients.

Anticipated Results: We anticipated that the ADHD group will have poorer time perception, particularly in difficult tasks, and the impairment will be reduced after treatment with medication

DETAILED DESCRIPTION:
BACKGROUND Children with attention-deficit/hyperactivity disorder (ADHD), a common, impairing neuropsychiatric disorder, are more likely to have difficulties planning and organizing. They cannot do things in an efficient way, cannot feel the limit of time schedule, and have difficulties awaiting their turns (Barkley, 1998). They often spend much longer time in homework, forget to accomplish routines or prescheduled work. Such behaviors often result in conflicts in the parent-child relationship.

In order to measure time perception, Barkley et al. (1997) developed two rating scales to evaluate children's sense of time and their ability of time management. They found an association between ADHD and poor time management. Barkley's (1998) comprehensive model suggested that time perception deficits in children with ADHD are due to deficits in behavioral inhibition and executive functions. Barkley et al's time reproduction tasks showed that children (1997), adolescents and young adults (2001) with ADHD had significantly more errors.

Recent studies focused on the associations of time reproduction with sustained attention, working memory, and behavioral inhibition. Kerns et al. (2001) reported a positive association between performance on a measure of attention (CPT) and a time reproduction task with a mixed result on the relationships between time reproduction and inhibitory control and working memory. McInerney and Kerns (2003) found the associations of time reproduction with working memory and behavioral inhibition, which lend support to the notion that time reproduction requires executive functions.

Smith et al. (2002) found that children with ADHD are more impaired in time discrimination threshold and less sensitive in fine time perception. This finding was later supported by Toplak et al (2003, 2005) using different modalities such as visual and auditory stimuli.

All the time perception tasks require the ability to allocate attention; however, different tasks involve other different mental abilities for estimation of duration of presentation of a target. Verbal estimation task is more related to the length of one's subject time unit, as synonymous inner clock speed. Time discrimination and time reproduction are related to the duration comparison. In addition to estimating the duration in the time discrimination task, subjects need to allocate their attention for a longer time and then to produce a target with the same duration by using some executive functions such as behavioral inhibition, sustain attention and working memory.

Few studies examined the efficacy of medication treatment of ADHD on time perception. Although Barkley et al., (1997) did not find effect of psychostimulants on the time reproduction, Baldwin et al. (2004) found that MPH significantly decrease time response variability, and decreased lever holds of extremely short durations. These findings suggest that administration of MPH resulted in more precise time performance without changing the mean duration of lever holds.

Although current empirical data from a few studies support that ADHD have time perception deficit and MPH may be effective in improving time reproduction, there is no information about time perception deficits in the Chinese population. In view of this, we will conduct a study to investigate the clinical and treatment aspects of time perception among children and adolescent with ADHD.

Specific Aims:

1. to examine the developmental and gender effect on the performance in time perception;
2. to explore the deficit in time estimation, time discrimination, and time reproduction in children and adolescents with ADHD as compared to normal controls;
3. to identify the association between ADHD symptoms and performance in time perception tasks; and
4. to investigate the efficacy of MPH on the time perception measures among children and adolescents with ADHD.

METHODS Participants We will recruit 100 patients with DSM-IV ADHD, aged 9 to 16 years, and 100 school controls. The 100 patients with ADHD will reassessed with time perception tasks 3 to 6 months later after treatment at outpatient department.

Measures

1. Diagnostic Tool Chinese version of Kiddie-Schedule for Affective Disorders and Schizophrenia- Epidemiology version (K- SADS-E) Development of the CK-SADS-E was carried out by the Child Psychiatry Research Group in Taiwan (Gau and Soong, 1999), which included a two-stage translation and modification of several items with psycholinguistic equivalents relevant to the Taiwanese culture. Previous studies have proved the CK-SADS-E to be a reliable and valid instrument to assess child psychiatric disorders in Taiwan. The CK-SADS-E has been widely used in a variety of studies on the mental illness of children and adolescents in Taiwan (e.g., Gau et al., 2005).
2. Questionnaires Chinese version of the Conners' Parent Rating Scale-Revised: Short Form (CPRS-R: S) A 27-item parent-reported rating scale for the assessment of behavioral symptoms, with four subscales: Oppositional (6 items), Inattention/Cognitive Problems (6 items), Hyperactivity/Impulsivity (6 items), and ADHD-index (12 items), was used. Each item is rated on a 4-point Likert scale-0 for not true at all (never, seldom), 1 for just a little true (occasionally), 2 for pretty much true (often, quite a bit), and 3 for very much true (very often, very frequent) (Gau et al., 2006).

   The Chinese version of the Conners' Teacher Rating Scale-Revised: Short Form (CTRS-R:S) A 28-item teacher-reported rating scale for the assessment of behavioral symptoms, with four subscales: Oppositional (5 items), Cognitive Problems/Inattention (5 items), Hyperactivity/Impulsivity (7 items), and ADHD-index (12 items), was used. Like the CPRS-R:S, each item is rated from 0 for not true at all (never, seldom) to 3 for very much true (very often, very frequent) (Gau et al., 2006).

   The Swanson, Nolan, and Pelham, version IV ( SNAP-IV Scale) The SNAP-IV is a 26-item rating scale consisting of the DSM-IV symptoms for the Inattention (Item 1-9) and the Hyperactivity/Impulsivity domains (Item 10-18) of the criteria for ADHD, and the oppositional symptoms (Item 19-26) of the criteria for ODD. Several studies have used different versions of the SNAP, either parent or teacher form, as an outcome measure to assess the efficacy of treatment for ADHD (e.g., Steele et al., 2006). Regarding psychometric properties of the SNAP rating scale, the Chinese version of SNAP-IV showed satisfactory test-retest reliability (intraclass correlation= 0.59~0.72), internal consistency (alpha=0.88~0.90), concurrent validity (Pearson correlations = 0.56~0.72), and discriminant validity (Liu et al., 2006).
3. Neuropsychological Tests Verbal Estimation Task This task, modified from Barkley et al. (2001a), is to assess the length of participant's subjective temporal unit. First, the green circle is present on the central for several seconds then it will disappear. Subject is asked the duration of each target in 5, 12, 17, and 25 seconds. For each presentation in random, there are two trials rendering eight trials in total.

Time Discrimination Task Time discrimination task, modified from Smith et al. (2002) presents the green circle on the left first, followed by the red circle on the right. The subject is asked to press the key to indicate the circle with longer duration. The standard stimuli and comparison last for 1000ms, and 1350ms, respectively. The two circles are randomly presented. If the answer is correct, the comparison duration decreases in 15ms; if the answer is wrong, the comparison duration increases in 15ms. The task continued either until the subject had made six reversals, or until 20 trials, whichever occurs first.

Time Reproduction Task The time reproduction task is modified from Barkley et al. (1997). First, the green circle is present on the central for seconds with five durations: 2, 5, 10, 12, and 17seconds. Subject is asked to press key to create the same temporal duration as green circle. Two trials are given at each of these five durations with random presentation.

The raw time reproduction is converted into the absolute discrepancy score, which consists of the absolute value of magnitude of the discrepancy between the participant's time production and the interval presented to the subject to measure the extent of errors.

Conners' Continuous Performance Test (CPT) The CPT requires tabbing on the space key when any character other than X shown on the screen. There were six sets in total, with 20 characters within each set. The Inter-Stimulus Intervals (ISIs) are 1, 2, and 4 seconds, and different ISIs varied between sets. Each character maintains on the screen for 250 ms. Correct hits, omission errors, commission errors, and reaction times will be collected as indices of response selection and capacity/focus. The d' value known as a discriminate factor is one of the indices for sustained attention.

The Wechsler Intelligence Scale for Children - the 3rd edition short form WISC-III (Wechsler, 1991) is a well established scale designed to assess the Full-Scale IQ (FSIQ) of children under age of 16. It includes 13 subtests to test children's cognitive ability of different dimensions. Test result is represented by Verbal IQ, Performance IQ, and Full-Scale IQ. The present research conducted a quad combination of WISC short form including subtests of Symbol Search, Arithmetic, Block Design, and Verbal. Previous research suggested the mentioned combination have good reliability (rxx = .91) and validity (rxx = .90) (Silverstein, 1982), and is preferred while conducting research to estimate FSIQ.

Procedure We will obtain written informed consent of all subjects from both children and their parents. The day prior to the date of receiving neuropsychological tasks, children will be asked to halt medication (if they are not drug-naïve patients) in order to obtain their test results as baseline data to make comparison with their performance after treatment with medication for 3 months or one year.

The testing procedure is as follows: (1) In addition to clinical diagnosis, subjects' mothers will receive K-SADS-E interview to make psychiatric diagnosis. (2) All subjects (ADHD group and normal controls) will be assessed IQ and a series of time perception tasks. Their parents will complete the SNAP-IV and CPRS-R:S and teachers will complete the CTRS-R:S. (3) After receiving medication for ADHD for 3 months and for one year, children will be reassessed by time perception tasks and CPT. Their parents and teachers will be asked to complete the same rating scales.

Anticipated Results:

We anticipated that the ADHD group will perform poorer in time estimation, time discrimination, and time reproduction, particularly in difficult tasks, and the impairment will be reduced after treatment with medication.

ELIGIBILITY:
Inclusion Criteria:

* Case group:

  * DSM-IV ADHD,
  * aged 9 to 16 years,
  * IQ > 80,
  * Subjects and Parents consent to the study.
* Control:

  * No ADHD,
  * aged 9 to 16 years,
  * IQ > 80,
  * Subjects and Parents consent to the study.

Exclusion Criteria:

* A history of brain injury or epilepsy,
* visual/auditory deficit or were diagnosed as having motor disorder,
* obsessive-compulsive disorder,
* mental retardation, and depression.
* In order to recruit a population of pure ADHD (without other psychiatric comorbidities), children who are comorbid with oppositional defiant disorder (ODD) or conduct disorder (CD) were excluded, though the concurrence of ODD/CD and ADHD

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with and without ADHD
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2006-05; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hwang SL, Gau SS, Hsu WY, Wu YY. Deficits in interval timing measured by the dual-task paradigm among children and adolescents with attention-deficit/hyperactivity disorder. J Child Psychol Psychiatry. 2010 Mar;51(3):223-32. doi: 10.1111/j.1469-7610.2009.02163.x. Epub 2009 Sep 15. PMID 19754502